CLINICAL TRIAL: NCT03088969
Title: Validation of the French Version of the Questionnaires of Self-efficacy Received From the People With a Chronic Low Back Pain After Return to the Work (10 and 19 Items)
Brief Title: Validation of the French Version RTWSE (Return To Work Self Efficacy Scale)
Acronym: RTWSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-309
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Function; Self-efficacy; Return to work; Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with a chronic back pain
  Interventions: Other: questionnaire RTWSE

INTERVENTIONS:
Other: questionnaire RTWSE — The evaluation of the self-efficiency perceived of return in the work of the patients by a validated auto-questionnaire is thus an additional objective parameter determining the risk factors of unfavorable evolution of the patients with Low Back Pain. This parameter also allows highlight other levers of actions in the therapeutic education.

SUMMARY:
The back pain connected to the work stay a major problem in industrialized countries, in particular because of the repercussions of this affection on the work (sick leave, absenteeism, handicap and inaptitude). It is difficult to consider among all the patients with a Chronic Low Back Pain in the work: how much they are going to stop. However, Investigator can consider that approximately 20 % of the patients have a sick leave. Several studies showed well that more the sick leave work stoppage goes on more the risk of not resumption of work increases. Several risk factors were associated to the evolutionary forecast of the pathology and thus to the extension extra time of the sick leave: individual, environmental, psychosocial and organizational.

The evaluation of the self-efficiency perceived of return in the work of the patients by a validated auto-questionnaire is thus an additional objective parameter determining the risk factors of unfavorable evolution of the patients with Low Back Pain. This parameter also allows highlight other levers of actions in the therapeutic education.

DETAILED DESCRIPTION:
First stage: the translation of the RTWSE in French followed the recommendations of the literature, which recommend a double translation, then a double back - translation with synthesis of the data in every stage. A final commission deliberate then a final translation, culturally adapted.

The second stage: the RTWSE is given to the patients with a Chronic Back Pain in the program of functional restoration of the rachis. Questionnaire FABQ, BARBECUE and Quebec are also given to the patient to obtain the status "faith" and the "functional" status. The questionnaire JDI as well as the analog visual scale is given to estimate the global professional satisfaction. The pain is estimated by a digital scale. The score IPAQ allows to estimate the level of physical activity of the patients. The HAD allows to estimate the level of anxiety and depression of the patients.

The additional questionnaires used for several reasons: in routine for the evaluation of the patients with a Chronic Back Pain; to characterize the patients and within the framework of the study for the validity of convergence and difference of questionnaires RTWSE 10 and 19 items.

The third stage: the questionnaire RTWSE is given again to the patient at 72 hours interval while the state of the patient is considered as stable.

The fourth stage: the questionnaires are given at J21 and in 2 months apart for the study of the sensibility in the change with the FABQ, BARBECUE, Quebec and the IPAQ.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Adult (>18 years old)
* Chronic Low Back Pain evolving for at least 3 months
* Acceptance to participate in the study
* Patients affiliated to a social security scheme (beneficiary entitled)

Exclusion Criteria:

* Patient under guardianship, or protection of justice.
* Patient in the incapacity to answer the questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a chronic back pain
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of the questionnaires RTWSE (Return To Work Self Efficacy Scale, 10 et 19 items) | at 0 day
Psychometric properties of the questionnaires RTWSE (Return To Work Self Efficacy Scale, 10 et 19 items) | at 3 days
Psychometric properties of the questionnaires RTWSE (Return To Work Self Efficacy Scale, 10 et 19 items) | at 21 days
Psychometric properties of the questionnaires RTWSE (Return To Work Self Efficacy Scale, 10 et 19 items) | at 2 months

SECONDARY OUTCOMES:
The fears and the faiths measured by questionnaire FABQ | at day 0
The fears and the faiths measured by questionnaire FABQ | at 21 days
The fears and the faiths measured by questionnaire FABQ | at 2 months
Average change from baselin in the pain intensity measured on a Visual Analogical Scale (VAS) | at day 0
Average change from baselin in the pain intensity measured on a Visual Analogical Scale (VAS) | at day 3
Average change from baselin in the pain intensity measured on a Visual Analogical Scale (VAS) | at day 21
Average change from baselin in the pain intensity measured on a Visual Analogical Scale (VAS) | at 2 months
Level of physical activity measured by short questionnaire IPAQ | at day 0
Level of physical activity measured by short questionnaire IPAQ | at 2 months
The 14-item Beliefs and Behaviors Questionnaire (BBQ) measures beliefs, experiences and adherent behavior related with Low Back pain | at day 0
The 14-item Beliefs and Behaviors Questionnaire (BBQ) measures beliefs, experiences and adherent behavior related with Low Back pain | at 3 days
The 14-item Beliefs and Behaviors Questionnaire (BBQ) measures beliefs, experiences and adherent behavior related with Low Back pain | at 2 months
The knowledge of emotional state measured by questionnaire HAD | at day 0
The knowledge of emotional state measured by questionnaire HAD | at 21 days
Self-assessment of the incapacity, that deals with the echo on the everyday life measured by questionnaire QUEBEC | at day 0
Self-assessment of the incapacity, that deals with the echo on the everyday life measured by questionnaire QUEBEC | at 21 days
Self-assessment of the incapacity, that deals with the echo on the everyday life measured by questionnaire QUEBEC | at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Rossignol M, Rozenberg S, Leclerc A. Epidemiology of low back pain: what's new? Joint Bone Spine. 2009 Dec;76(6):608-13. doi: 10.1016/j.jbspin.2009.07.003. No abstract available. PMID 19818666
- [Background] Gourmelen J, Chastang JF, Ozguler A, Lanoe JL, Ravaud JF, Leclerc A. Frequency of low back pain among men and women aged 30 to 64 years in France. Results of two national surveys. Ann Readapt Med Phys. 2007 Nov;50(8):640-4, 633-9. doi: 10.1016/j.annrmp.2007.05.009. Epub 2007 Jun 27. English, French. PMID 17631977
- [Background] Ozguler A, Leclerc A, Landre MF, Pietri-Taleb F, Niedhammer I. Individual and occupational determinants of low back pain according to various definitions of low back pain. J Epidemiol Community Health. 2000 Mar;54(3):215-20. doi: 10.1136/jech.54.3.215. PMID 10746116
- [Background] Brouwer S, Franche RL, Hogg-Johnson S, Lee H, Krause N, Shaw WS. Return-to-work self-efficacy: development and validation of a scale in claimants with musculoskeletal disorders. J Occup Rehabil. 2011 Jun;21(2):244-58. doi: 10.1007/s10926-010-9262-4. PMID 20865445
- [Background] Shaw WS, Reme SE, Linton SJ, Huang YH, Pransky G. 3rd place, PREMUS best paper competition: development of the return-to-work self-efficacy (RTWSE-19) questionnaire--psychometric properties and predictive validity. Scand J Work Environ Health. 2011 Mar;37(2):109-19. doi: 10.5271/sjweh.3139. Epub 2011 Jan 4. PMID 21203742
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752